CLINICAL TRIAL: NCT01905267
Title: Mindfulness Intervention to Study the Neurobiology of Depression
Acronym: MIND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Rachel Jacobs, Research Assistant Professor, Licensed Clinical Psychologist, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2012-0689
Record Dates: First submitted 2013-07-10; First posted 2013-07-23 (Estimated); Results first posted 2018-07-30 (Actual); Last update posted 2018-07-30 (Actual); Status verified 2017-10

CONDITIONS: Depression
Keywords: mindfulness; relapse prevention; recovery; depression; adolescents
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Experimental): Participants randomized to the experimental condition will receive 8 weeks of individual treatment with Rumination-Focused Cognitive Behavior Therapy
  Interventions: Behavioral: Rumination-Focused Cognitive Behavior Therapy
- Control (No Intervention): Participants randomized to the control arm will complete questionnaires and receive mood monitoring for the duration of the study

INTERVENTIONS:
Behavioral: Rumination-Focused Cognitive Behavior Therapy — This intervention targets rumination and other maladaptive forms of emotion regulation such as suppression and avoidance and provides skills training in effective coping strategies. Mindfulness is a key component of this intervention as a strategy for disengaging from one's thoughts. Strategies from Dialectical Behavior Therapy (DBT), such as the use of effective interpersonal skills, are also included as methods for regulating strong emotion. Rumination-Focused Cognitive Behavior Therapy is a structured, manual based program designed to be delivered weekly over eight weeks. Sessions are 60-90 minutes in length.
  Arms: Treatment

SUMMARY:
The Pediatric Mood Disorders Program at the University of Illinois at Chicago is conducting a research study examining how mindfulness can help teenagers stay healthy and prevent depression relapse.

DETAILED DESCRIPTION:
Study involves:

* Brain scan using fMRI technology
* Questions about mood and behavior
* Meeting with a clinician
* Possibility of 8 weekly treatment sessions using mindfulness
* Ongoing assessment of depression for next 2 years

Eligible participants will be compensated for their time.

ELIGIBILITY:
Inclusion Criteria:

* between the ages of 12 and 18
* history of major depressive disorder

Exclusion Criteria:

* braces
* afraid of small spaces

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 33 (Actual)
Dates: Start 2013-03; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel H Jacobs, PhD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago Pediatric Mood Disorders Program, Chicago, Illinois, United States

REFERENCES:
- [Derived] Bessette KL, Jacobs RH, Heleniak C, Peters AT, Welsh RC, Watkins ER, Langenecker SA. Malleability of rumination: An exploratory model of CBT-based plasticity and long-term reduced risk for depressive relapse among youth from a pilot randomized clinical trial. PLoS One. 2020 Jun 17;15(6):e0233539. doi: 10.1371/journal.pone.0233539. eCollection 2020. PMID 32555582
- [Derived] Jacobs RH, Watkins ER, Peters AT, Feldhaus CG, Barba A, Carbray J, Langenecker SA. Targeting Ruminative Thinking in Adolescents at Risk for Depressive Relapse: Rumination-Focused Cognitive Behavior Therapy in a Pilot Randomized Controlled Trial with Resting State fMRI. PLoS One. 2016 Nov 23;11(11):e0163952. doi: 10.1371/journal.pone.0163952. eCollection 2016. PMID 27880789

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment | Control
Started | 17 | 16
Completed | 15 | 14
Not Completed | 2 | 2
Not completed — Physician Decision | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment | Control | Total
Number analyzed (Participants) | 17 | 16 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.41 (1.97) | 15.69 (1.89) | 15.55 (1.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 19
  Male | 8 | 6 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 4 | 8
  White | 8 | 9 | 17
  More than one race | 4 | 2 | 6
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Children's Depression Rating Scale - Revised
Description: clinician measure completed with adolescent and parent Total scores reported. Range is between 17-119 Higher scores mean higher depressive symptoms
Time Frame: Baseline, 8 week
Population: completers sample
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment | Control
Number analyzed (Participants) | 15 | 14
units on a scale
  Baseline | 27.47 (3.94) | 28.00 (6.82)
  8 week | 25.53 (4.22) | 31.86 (10.99)

2. Secondary Outcome: Change in Reynolds Adolescent Depression Scale
Description: Self report adolescent depression total score. Range is 30-120 with higher scores meaning greater depressive symptoms.
Time Frame: Baseline, 8 week
Population: 8 week completers sample
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment | Control
Number analyzed (Participants) | 15 | 14
units on a scale
  Baseline | 64.41 (12.12) | 63.50 (12.42)
  Week 8 | 56.93 (13.22) | 61.5 (13.77)

ADVERSE EVENTS:
Time Frame: two years following 8 week intervention period every six months
Description: Study staff informed of hospitalizations for suicidality or increasing depressive symptoms during course of KSADS clinical assessments
Arm/Group | Treatment | Control
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/17 | 5/16
Other Adverse Events (participants affected / at risk) | 0/17 | 0/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=17) | Control (N=16)
Suicidality (Psychiatric disorders) | 0 (0) | 5 (5) — Five participants were hospitalized for suicidality or suicidal gestures.

LIMITATIONS AND CAVEATS:
Small number of subjects

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Informed Consent Form (2014-07-31): https://cdn.clinicaltrials.gov/large-docs/67/NCT01905267/ICF_000.pdf
  • Study Protocol (2014-06-30): https://cdn.clinicaltrials.gov/large-docs/67/NCT01905267/Prot_001.pdf
  • Statistical Analysis Plan (2014-07-01): https://cdn.clinicaltrials.gov/large-docs/67/NCT01905267/SAP_002.pdf